CLINICAL TRIAL: NCT02404207
Title: The Effect of High-Oleic Soybean Oil on Biomarkers of Risk for Metabolic Syndrome
Brief Title: Soybean Oil Trial of cArdiovascular Risk
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Baer, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HS50
Record Dates: First submitted 2015-03-18; First posted 2015-03-31 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Disease; Diabetes; Metabolic Syndrome
Keywords: Prevention
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Metabolic Syndrome | interventions — Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Soybean oil (Active Comparator)
  Interventions: Other: Soybean oil
- High-oleic soybean oil (Experimental)
  Interventions: Other: High-oleic soybean oil
- High-oleic soybean oil + fully hydrogenated soybean oil (Experimental)
  Interventions: Other: High-oleic soybean oil + fully hydrogenated soybean oil
- Palm olein + palm stearin (Active Comparator)
  Interventions: Other: Palm olein + palm stearin

INTERVENTIONS:
Other: Soybean oil — Participants will be fed soybean oil as part of a controlled (typical American) diet.
  Arms: Soybean oil
Other: High-oleic soybean oil — Participants will be fed high-oleic soybean oil as part of a controlled (typical American) diet.
  Arms: High-oleic soybean oil
Other: High-oleic soybean oil + fully hydrogenated soybean oil — Participants will be fed a blend of high-oleic soybean oil and fully hydrogenated soybean oil as part of a controlled (typical American) diet.
  Arms: High-oleic soybean oil + fully hydrogenated soybean oil
Other: Palm olein + palm stearin — Participants will be fed a blend of palm olein + palm stearin as part of a controlled (typical American) diet.
  Arms: Palm olein + palm stearin

SUMMARY:
The study will determine the effects of different types of soybean oils on biomarkers of risk for cardiovascular disease and diabetes. There will be four 4-week diet periods in which participants will consume the following oils, within the context of a controlled diet: soybean oil, high-oleic soybean oil, blend of high oleic soybean oil & fully hydrogenated soybean oil, and blend of palm olein & palm stearin.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 70 years at beginning of study
* LDL-cholesterol between 120 and 160 mg/dl
* Less than 2+ risk factors for coronary heart disease (risk factors include: blood pressure > 140/90 mm Hg or on blood pressure medication; HDL-cholesterol < 40 mg/dl; age greater than 45 yrs for males & greater than 55 yrs for females; family history of premature coronary heart disease (CHD in male first degree relative <55 years; CHD in female first degree relative <65 years)

Exclusion Criteria:

* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Use of prescription or over-the-counter medications or supplements that alter lipid metabolism.
* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of bariatric or certain other surgeries related to weight control
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanolamine, ephedrine, caffeine) during and for at least 6 months prior to the start of the study or a history of a surgical intervention for obesity
* Unwillingness to abstain from herbal supplements for two weeks prior to the study and during the study
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Known (self-reported) allergy or adverse reaction to study foods
* Active cardiovascular disease (such as a heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within the last three months, stroke, or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in the past six months)
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in lipid profile | At baseline and end of each 4-week diet period
  Lipids and lipoproteins, such as total cholesterol, LDL-cholesterol, HDL-cholesterol, triacylglycerides, Apo AI, ApoAII, ApoB, apolipoprotein size, and cholesterol ester composition, will be measured in the blood.

SECONDARY OUTCOMES:
Change in systemic inflammation | At baseline and end of each 4-week diet period
  Markers of systemic inflammation will be measured, such as IL-6, CRP, and isoprostanes.
Change in hemostasis | At baseline and end of each 4-week diet period
  Markers of hemostasis will be measured, such as fibrinogen and factor VIIc.
Change in oxidation | At baseline and end of each 4-week diet period
  Markers of oxidation will be measured, such as 4-hydroxynonenal, vitamin E, oxidized LDL, lipid hydroperoxides, and malondialdehyde.
Change in vascular health | At baseline and end of each 4-week diet period
  Markers of vascular health will be measured, such as ICAM, VCAM, eSelectin, and blood pressure.
Change in glucose | At baseline and end of each 4-week diet period
  Fasting blood glucose will be measured.
Change in insulin | At baseline and end of each 4-week diet period
  Fasting insulin will be measured.
Change in body composition | At baseline and end of each 4-week diet period
  Dual-energy x-ray absorptiometry (DEXA; fat and lean mass, visceral fat) will be measured.
Change in waist circumference | At baseline and end of each 4-week diet period

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States